CLINICAL TRIAL: NCT02168387
Title: Efficacy of Percussive Ventilation Therapy (MetaNeb ®) Compared With Mucolytic Agents for Atelectasis in the Mechanically Ventilated Pediatric Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00026503
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Atelectasis
Keywords: atelectasis; continuous high frequency oscillator; acetylcysteine; dornase alfa
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Acetylcysteine; dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous high frequency oscillator (CHFO) (Active Comparator): Subjects randomized to receive therapy with the CHFO will receive a 20 minute treatment every 6 hours for 48 hours.
  Interventions: Device: continuous high frequency oscillator (CHFO)
- medication (Active Comparator): Subjects randomized to receive the medications will receive acetylcysteine and dornase alfa, two medications frequently used in the treatment of atelectasis. The medications will alternate every 6 hours for 48 hours.
  Interventions: Drug: Acetylcysteine; Drug: dornase alfa

INTERVENTIONS:
Device: continuous high frequency oscillator (CHFO)
  Arms: continuous high frequency oscillator (CHFO)
Drug: Acetylcysteine
  Arms: medication
Drug: dornase alfa
  Arms: medication

SUMMARY:
The purpose of this study is to evaluate whether a therapy that uses a machine called a continuous high frequency oscillator (CHFO) is more successful at removing mucus than medications that thin out the mucus.

DETAILED DESCRIPTION:
Both of these therapies (CHFO and medication) are currently used in the Pediatric Intensive Care Unit and Pediatric Cardiac Intensive Care Unit. This research study is being done because the investigator is trying to learn if the mechanical removal of mucus with CHFO will effectively re-inflate the collapsed area of lung. Specifically, the study team will determine if CHFO can improve lung inflation with the same or improved vital signs (heart rate, blood pressure, and breathing rate), and the same or improved ability to help the lungs move oxygen into the blood.

One of the problems with the medication approach is that while it thins out the mucus, actual removal from the lung requires a strong cough which is difficult for infants and children to produce when they are sedated and on a ventilator (breathing machine).

Thus, the aim of this research study is to test whether children with atelectasis on a ventilator are more likely to improve with mechanical removal of their mucus with the CHFO as compared with medications that thin out the mucus. CHFO and all the medications used in this study are part of the standard of care for atelectesis. However, there is no information on which combination works best and no one agrees that one approach is more effective than another. Usually patients are evaluated for 48 hours after starting treatment, before adding or making any changes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from parent or legal guardian.
2. Age < 18 years and admitted to the PICU or PCICU.
3. Conventionally ventilated.
4. Mucolytics are being initiated by clinical team for treatment of atelectasis.
5. Endotracheal tube ≥ 3.5 mm internal diameter.

Exclusion Criteria:

1. Receiving chronic mucolytic or continuous high frequency oscillation therapy.
2. Clinically significant pleural effusion.
3. Status post cardiothoracic surgery with open chest.
4. Pneumothorax.
5. Pulmonary hemorrhage.
6. Escalating doses of vasoactive agents (i.e. dopamine or epinephrine).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Cheifetz, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All mechanically ventilated patients 0-17 years of age admitted to the Pediatric Intensive Care Unit (PICU) and Pediatric Cardiac Intensive Care Unit (PCICU) from January 2011 to March 2012 with radiographic evidence of atelectasis for which mucolytics or CHFO therapy were being initiated by the patient care team were screened for enrollment.
Groups:
- Medication: Subjects randomized to receive the medications will receive acetylcysteine and dornase alfa, two medications frequently used in the treatment of atelectasis. The medications will alternate every 6 hours for 48 hours.
  Acetylcysteine
  dornase alfa
- Continuous High Frequency Oscillator (CHFO): Subjects randomized to receive therapy with the CHFO will receive a 20 minute treatment every 6 hours for 48 hours.
  continuous high frequency oscillator (CHFO)
Period: Overall Study
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO)
Started | 20 | 19
Completed | 13 | 16
Not Completed | 7 | 3
Not completed — Planned exubation | 6 | 3
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO) | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Customized [Number; unit: participants]
  less than or equal to 1 year | 11 | 10 | 21
  greater than 1 year | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Atelectasis
Description: An atelectasis score (AS), as published by Deakins, et al. 2002, was assigned to each radiograph as follows:
  0 Complete resolution of collapse
  1. Partial collapse of 1 segment or lobe
  2. Partial collapse of ≥ 2 segments or lobes
  3. Complete collapse of 1 segment or lobe
  4. Complete collapse of ≥ 2 segments or lobes
  In the event of inter-rater disagreement, the scores were averaged. Improvement was defined as any decrease in AS ≥ 0.5. Worsening was defined as an increase in AS ≥ 0.5 or escalation of respiratory support modality (i.e. high frequency ventilation).
Time Frame: after 48 hours of therapy
Measure: Number; unit: participants
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO)
Number analyzed (Participants) | 13 | 16
participants
  Improved in 48 h | 6 | 7
  Worse in 48 hr | 3 | 6
  No change in 48 hr | 4 | 3

2. Secondary Outcome: Change in Capnography (Vd/Vt)
Description: The deadspace-to-tidal volume (Vd/Vt) ratio is a parameter that is measured in mechanically ventilated patients as a way to assess the severity of gas exchange impairment and to assist in determining whether a patient is ready to be weaned from the ventilator. The change from baseline was measured at 48 hours, with a decreasing ratio indicating improvement.
Time Frame: baseline and 48 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO)
Number analyzed (Participants) | 13 | 16
ratio | -0.04 (0.08) | 0.03 (0.09)

3. Secondary Outcome: Change in Quantity and Quality of Suctioned Mucus
Time Frame: baseline and 48 hours
Population: These data were not obtained due to technical difficulties.
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Medication | Continuous High Frequency Oscillator (CHFO)
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication (N=20) | Continuous High Frequency Oscillator (CHFO) (N=19)
death due to underlying disease (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size in a single center study. Children who were extubated prior to the end of the study were not accounted for, as this was not a primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes